CLINICAL TRIAL: NCT00516945
Title: A Randomized Controlled Study Comparing the Impact of Prophylactic Versus Deferred Lamivudine on the Delivery of Cytotoxic Chemotherapy in Hepatitis B Surface-antigen Positive Patients With Malignant Solid Tumor
Brief Title: A Study to Investigate Whether the Immediate Use or Deferred Use of an Anti-viral Drug Lamivudine Will Help to Better Safe-guard the Delivery of Chemotherapy in Patients With Cancer Who Are Also Hepatitis B Carriers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KC/KE04-0046/FR-2; HARECCTR0500016
Record Dates: First submitted 2007-08-15; First posted 2007-08-16 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-07

CONDITIONS: Hepatitis B; Neoplasms
Keywords: hepatitis B during cancer chemotherapy
MeSH Terms: conditions — Hepatitis B; Neoplasms | interventions — Lamivudine

INTERVENTIONS:
Drug: Lamivudine

SUMMARY:
Patients with non-lymphoma and non-leukaemia cancer who are also hepatitis B carriers will have a risk of hepatitis B reactivation during chemotherapy. Lamivudine can be used effectively to control hepatitis upon reactivation during chemotherapy and the chemotherapy may not need to be interrupted. The study aims to investigate whether adding the anti-viral drug Lamivudine at the start of chemotherapy for all patients, rather than at the time of hepatitis reactivation for those with reactivation, will help to improve the delivery of chemotherapy in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with histology-proven malignant solid tumor other than malignant lymphoma
2. Patients with age between 18 and 75
3. Patients with Karnofsky performance score (KPS) of at least 60
4. Patients planned for at least 4 cycles of intensive cytotoxic chemotherapy (either as part of curative therapy or as palliative therapy), except for those receiving single agent cisplatin chemotherapy alone concurrently with radiation for radiosensitization
5. Patients with at least 6 months' life expectany from date of recruitment
6. Patients with normal liver function tests including alanine aminpotransferase (ALT), alkaline phosphatase (ALP), gamma glutamyl-transpeptidase (GGT), and bilirubin
7. Patients with no known history of radiological &/or histological diagnosis of chronic active hepatitis or cirrhosis of any cuase, or history of prior hepatitis B reactivation, or prior chronic therapy for HBV within 6 months
8. Patients with no evidence of autoimmune hepatitis, hepatitis C or delta virus infection, HIV infection or radiological evidence of liver metastasis
9. Patients with negative pregnancy test for female gender of child-bearing age

Exclusion Criteria:

1. Patients with age < 18 and > 75
2. Patients with Karnofsky performance score (KPS) of < 60
3. Patients planned for single agent cisplatin chemotherapy alone concurrently with radiation for radiosensitization
4. Patients with < 6 months' life expectancy from date of recruitment
5. Patients with abnormal liver function tests including alanine aminotransferase (ALT), alkaline phosphatase (ALP), gamma glutamyl- transpeptidase (GGT), and bilirubin
6. Patients with known history or radiological and/or histological diagnosis of chronic active hepatitis or cirrhosis of any cause, or history of prior hepatitis B reactivation, or prior chronic therapy for HBV within 6 months
7. Patients with autoimmune hepatitis, hepatitis C or delta virus infection, HIV infection or radiological evidence of liver metastasis
8. pregnant female patients

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2004-09; Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
incidence of chemotherapy interruptions | during chemotherapy of the study period

SECONDARY OUTCOMES:
incidence of and survival free from hepatitis B reactivation | during and after chemotherapy of the study period
HBeAg positive seroconversion and YMDD mutant development rates | during study period after chemotherapy
chemotherapy dose intensity reduction due to hepatitis B reactivation | during chemotherapy of the study period

CONTACTS AND LOCATIONS:
Overall Officials: Roger K C Ngan, Dr, Principal Investigator — Department of Clinical Oncology, Queen Elizabeth Hospital
Locations (1):
- Queen Elizabeth Hospital, Hong Kong, China